CLINICAL TRIAL: NCT00863239
Title: Phase 2B, Partially Blinded, Randomized Study in Treatment Naive HCV G1 to Compare the Efficacy, Safety, and Tolerability of Three Doses of Locteron Plus Ribavirin Given Bi-weekly in Comparison With PEG-Intron Plus Ribavirin Given Weekly
Brief Title: Phase 2B Dose Ranging Study of Locteron Plus Ribavirin to Treat HCV
Acronym: SELECT-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biolex Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BLX883-203
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Hepatitis C, Chronic
Keywords: treatment naive; genotype 1
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; locteron; polyethylene oxide-polybutylene terephthalate copolymer; peginterferon alfa-2b

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Locteron™ (controlled-release interferon alpha 2b) 320 µg as biweekly subcutaneous injection
  Interventions: Drug: ribavirin; Drug: Locteron™ (controlled-release interferon alpha 2b)
- 2 (Experimental): Locteron™ (controlled-release interferon alpha 2b) 480 µg as biweekly subcutaneous injection
  Interventions: Drug: ribavirin; Drug: Locteron™ (controlled-release interferon alpha 2b)
- 3 (Experimental): Locteron™ (controlled-release interferon alpha 2b) 640 µg as biweekly subcutaneous injection
  Interventions: Drug: ribavirin; Drug: Locteron™ (controlled-release interferon alpha 2b)
- 4 (Active Comparator): PEG-Intron™ (12 kDalton pegylated interferon alpha 2b) 1.5 µg/kg body weight weekly subcutaneous injection
  Interventions: Drug: ribavirin; Drug: PEG-Intron™

INTERVENTIONS:
Drug: ribavirin — Co-administered in all arms: oral ribavirin, 200 mg capsules. Subjects with body weight < 65 kg: 800 mg/day; Subjects with body weight 65-85 kg: 1000 mg/day; Subjects with body weight > 85 kg: 1200 mg/day.
  Other Names: Ribasphere®
Drug: Locteron™ (controlled-release interferon alpha 2b) — investigational controlled-release recombinant interferon alpha 2b formulated in 1500/77/23 PolyActive microspheres as a lyophilized powder, reconstituted with carboxymethyl cellulose immediately before subcutaneous injection every other week as part of the treatment of chronic hepatitis C
  Other Names: Locteron; PolyActive; BLX-883
  Arms: 1; 2; 3
Drug: PEG-Intron™ — commercially available pegylated interferon alpha 2b injected subcutaneously weekly in a dose of 1.5 ug/kg as part of the treatment of chronic hepatitis C
  Other Names: 12 kDalton pegylated interferon
  Arms: 4

SUMMARY:
The purpose of the study was to assess in subjects with chronic hepatitis C (treatment-naïve, genotype 1) receiving weight-based doses of ribavirin the virologic response to 3 dose levels of Locteron™, dosed every 2 weeks, in comparison with PEG-Intron™ dosed weekly.

DETAILED DESCRIPTION:
The aim of SELECT-2 study was to compare the safety and efficacy of Locteron to PegIntron. SELECT-2 was a 72-week Phase 2b, multicenter, international trial of treatment-naïve genotype-1 chronic HCV subjects who were randomized 1:1:1:1 and dosed with one of three doses [640ug (n=29), 480ug (n=29), 320ug (n=28)] of q2week Locteron or weekly doses of 1.5ug/kg PEG2b (n=30). Subjects received these regimens in combination with weight-based ribavirin (800-1400 mg) for up to 48 weeks. Subjects and staff were blinded to Locteron dose for the first 12 weeks. Subjects without early virologic response by 12 weeks, and without viral negativity by 24 weeks, discontinued treatment for lack of efficacy. Adverse events including flu symptoms and depression, Beck Depression Inventory (BDI), Short Form-36, HCV RNA and safety labs were measured at standard intervals at clinic visits through Week 72. In addition, daily subject self-reports of flu symptoms using an electronic subject reporting tool (ePRO) were collected for the first 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 through 69 years of age, inclusive
* Chronic hepatitis C genotype 1
* HCV ribonucleic acid (RNA) level > 10,000 IU/mL (by RT-PCR) at screening
* Creatine clearance ≥ 50 mL/min
* Neutrophil count > 1500 cells/mm3
* Platelet count > 90,000/mm3
* Hemoglobin > 12 g/dL for females and > 13 g/dL for males
* Female subjects of child-bearing potential agreeing to use dual methods for contraception
* Male subjects with female sexual partners agreeing to use effective birth control methods
* Negative serum pregnancy test for women of child-bearing potential • Compensated liver disease defined as INR < 1.5, conjugated bilirubin < 1.5 X ULN, serum albumin > 3.0 g/dL.

Exclusion Criteria:

* Prior antiviral treatment for hepatitis C
* Co-infection with HIV or hepatitis B virus
* Subjects with a body mass index (BMI) above 32 kg/m2
* Current or prior history of clinical hepatic decompensation
* Evidence of HCC
* Uncontrolled diabetes mellitus as evidenced by HbA1C ≥ 8.5% at screening
* Known hypersensitivity to interferon alfa or ribavirin
* Chronic liver disease other than HCV not limited to HBV, hemochromatosis, auto-immune hepatitis, alcoholic liver disease, non-alcoholic fatty liver disease)
* Clinically significant hemoglobinopathy such as thalassemia major and sickle cell anemia
* History of moderate, severe or uncontrolled psychiatric disease including depression and prior suicide attempts
* History of immune-mediated disease
* Significant renal or neurological disease
* Severe degree (> GOLD stage III) of chronic pulmonary disease (COPD) or active, severe asthma
* Subjects with severe cardiac disease (e.g., heart failure, recent [i.e., within 6 months prior to first dosing] myocardial infarction, angina, serious arrhythmias, including prolonged QTc [> 450 mSec], uncontrolled hypertension)
* History of significant central nervous system (including CNS trauma) or seizure disorders
* Cancer within the last 5 years, or previous cancer with a high risk of recurrence, including metastatic breast cancer; non-melanoma skin cancer is not an exclusion criterion
* History of solid organ or bone marrow transplantation
* Clinical or laboratory evidence of uncontrolled thyroid disease, e.g., by thyroid stimulating hormone (TSH) level > 1.2 X upper limit of normal
* Clinically significant retinopathy; this needs to have been excluded by an eye exam performed by an ophthalmologist within the last 6 months prior to screening for subjects with hypertension or diabetes mellitus
* Drug abuse or alcohol consumption within the last 6 months which, in the opinion of the investigator, may affect study participation or outcome. Subjects in a supervised methadone treatment program on a stable regimen for > 6 months may be considered
* Taken any experimental agent within 12 weeks prior to screening
* More than 30 days of systemic immunosuppressive medication to include steroids in doses equivalent to or greater than 10 mg prednisone per day within 30 days prior to screening (inhaled corticosteroids are allowed)
* Nursing mother or male partner of pregnant female.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2009-03; Primary Completion 2010-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
EVR: the proportion of subjects in each arm that have at least a 2 log drop in HCV RNA from Baseline | 12 weeks

SECONDARY OUTCOMES:
SVR: the proportion of subjects in each arm demonstrating HCV RNA undetectable (< 10 IU/mL) at the end of the follow-up period | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Walker A. Long, MD, Study Director — Biolex Therapeutics
Locations (24):
- United States (13):
  - eStudy site, Chula Vista, California
  - eStudy Site, Oceanside, California
  - Medical Associates Research Group, San Diego, California
  - University of Louisville Health Care Outpatient Center, Louisville, Kentucky
  - Maryland Digestive Disease Research, LLC, Laurel, Maryland
  - St. Louis University, St Louis, Missouri
  - AGA Clinical Research Associates, LLC., Egg Harbor, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Consultants for Clinical Research, Cincinnati, Ohio
  - The Liver Institute at Methodist Dallas, Dallas, Texas
  - Alamo Medical Center, San Antonio, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - McGuire DVAMC, Richmond, Virginia
- Bulgaria (7):
  - Tokuda Hospital, Sofia
  - UMHAT "Alexandrovska", Sofia
  - UMHAT "St Ivan Rilski", Sofia
  - UMHAT "Queen Giovanna - ISUL" EAD, Sofia
  - Medical Institute Ministry of Interior, Sofia
  - Military Medical Academy, Sofia
  - UMHAT "St Marina", Varna
- Fundacion de Investigacion de Diego, Santurce, Puerto Rico
- Romania (3):
  - Institute of Infectious Diseases, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - "Victor Babes" Clinical Hospital Craiova, Craiova

REFERENCES:
- [Result] 1. Lawitz E, Younossi Z, Mehra P, Rigney A, Krastev Z, Tchernev K, Takov D, Long WA. Early viral response of controlled-release interferon alpha2b and ribavirin vs. pegylated interferon alpha 2b and ribavirin in treatment-naïve genotype1 hepatitis C: 12 week results (SELECT-2 Trial). J Hepatology 52:S114 (abstract 272), 2010. (Presented to 45th Annual Meeting of the European Association for the Study of the Liver, April 15, 2010, Vienna, Austria.) 2. Long WA, Younossi Z, Lawitz E, Kotsev I, Takov D, Tchernev K, Rigney A, Ghalib R, Stoinov S, Balabanska R, Mehra P, Krastev Z. Timing and frequency of depression during HCV-treatment with controlled-release INFa2b (CR2b) vs. pegylated IFNa2b (PEG2b): Results from SELECT-2, a randomized open-label 72-week comparison in 116 treatment-naïve subjects with genotype-1 HCV. J Hepatology 54:S181-182, 2011 (abstract 446). (Presented to the 46th Annual Meeting of the European Association For The Study Of The Liver, Berlin, Germany, March 31, 2011.) 3. Lawitz E, Younossi Z, Mehra P, Rigney A, Krastev Z, Tchernev K, Takov D, Long WA. SVR for controlled-release interferon alpha-2b (CR2b) + ribavirin compared to pegylated intereferon alpha-2b + ribavirin in treatment-naïve genotype-1 (G1) hepatitis C: final results from SELECT-2. J Hepatology 54:S180-181, 2011 (abstract 444). (Presented to the 46th Annual Meeting of the European Association For The Study Of The Liver, Berlin, Germany, March 31, 2011.) 4. Younossi ZM, Lawitz EJ, Krastev Z, Rigney A, Tchernev K, Takov D, Ghalib RH, Long WA. SELECT-2 clinical trial assessing the efficacy and safety of controlled-release interferon alpha-2b (CR2b) +ribavirin (RBV) versus pegylated interferon alpha-2b (PEG2b) +RBV in treatment-naïve genotype-1 (G1) hepatitis C. Gastroenterology 140:S-942, 2011 (abstract su1868). (Presented to Digestive Disease Week 2011, Chicago, Illinois, May 8, 2011.)